CLINICAL TRIAL: NCT03672344
Title: Computer-based Social Skills Training for Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioStream Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08012018A
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Lookware TM (Active Comparator): Lookware TM computer-based video game that requires the subject to engage in social skills related exercises during simulated social interactions with game characters.
  Interventions: Device: Lookware TM
- Lookware TM Control Module (Placebo Comparator): Lookware TM Control Module is a version of the Lookware TM computer-based video game that excludes the social skills related exercises.
  Interventions: Device: Lookware TM Control Module

INTERVENTIONS:
Device: Lookware TM — Lookware TM is a computer-based video game that requires the subject engage in social skills related exercises that include certain visual behaviors. These exercises combine techniques from applied behavior analysis (ABA) and use of gaze-contingent eye tracking technology during simulated social interactions with 3D animated characters to target certain social skills deficits in children with autism spectrum disorder (ASD). The game is delivered through a laptop computer, eye tracker, and game controller.
  Arms: Lookware TM
Device: Lookware TM Control Module — Lookware TM Control Module is a version of the Lookware TM computer-based video game that excludes the social skills related exercises. The game is delivered through a laptop computer, eye tracker, and game controller.
  Arms: Lookware TM Control Module

SUMMARY:
The primary objective of this study is to evaluate changes in subject performance on social skills assessments after engaging in a gaze-controlled video game that leverages ABA principles of learning, in comparison to an alternative game. The secondary objectives of this study are to evaluate changes in subject gaze patterns during social skills assessments after engaging in the video game, including in comparison to an alternative game and to evaluate possible correlations in changes in social skills assessments with changes in subject game play performance.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 4-14.
2. Meets diagnostic criteria for ASD.
3. Estimated intelligence standard score of at least 40 (can be substituted for a receptive language score such as PPVT or use of the Differential Ability Scales, 2nd Edition (DAS-II)).
4. Parent reports difficulty with at least one of two social skills (via modified questions from the Social Responsiveness Scale)
5. English as the child's primary/first language (key measures used in the study do not have alternate language versions).
6. Attains a score equal to or less than 75% correct on the Ekman 60 Faces Test
7. The parent who completes the questionnaires needs to be proficient in English.
8. Has successfully played a video game using a Microsoft Xbox game controller, Sony PlayStation game controller, or other comparable game controller.
9. Parental/guardian permission (informed consent) and if appropriate, child assent.
10. Wi-Fi internet connection at subject's home/school/therapy center/research organization available for use by study laptop computer.

Exclusion Criteria:

1. History of seizures.
2. History of traumatic brain injury or other significant medical or neurological abnormality affecting motor or higher cortical functioning.
3. Certain visual, auditory, DSM 5, or conduct disorders (see below).
4. A visual disorder that cannot be corrected through the use of corrective lenses to a level of 20-40 in both eyes.
5. Use of corrective visual lenses that would significantly impede the valid collection of visual attention and gaze pattern data during dyadic interaction tasks.
6. Auditory impairment (that cannot be corrected by a hearing aid) that would significantly impede the valid collection of test measures.
7. Profound intellectual disability or sensory-motor difficulties that would preclude valid use of diagnostic instruments and/or use of a computer or mobile computing device.
8. A DSM 5 disorder or other psychiatric symptoms that would interfere with the participant's ability to participate in the study (e.g., active psychosis), per parent report.
9. History of one or more psychiatric hospitalizations.
10. Presence of significant symptoms of a conduct disorder.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Milestones Behavioral Services, Orange, Connecticut
  - Els for Autism Foundation, Jupiter, Florida
  - Positive Behavior Supports Corporation, Melbourne, Florida
  - Positive Behavior Supports Corporation, Miami, Florida
  - Positive Behavior Supports Corporation, West Palm Beach, Florida
  - Nashoba Learning Group, Inc., Bedford, Massachusetts
  - Y.A.L.E. School, Cherry Hill, New Jersey
  - Connect Plus Therapy, Inc., Cherry Hill, New Jersey
  - Partners in Learning, Inc., Clementon, New Jersey
  - Mary E. Keefe, Point Pleasant Beach, New Jersey
  - The Pathway School, Jeffersonville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No individuals who were enrolled in the study were subsequently excluded from the study.
Period: Overall Study
Arm/Group | Lookware TM | Lookware TM Control Module
Started | 25 | 29
Completed | 25 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lookware TM | Lookware TM Control Module | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.88 (2.37) | 9.14 (3.11) | 8.56 (2.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 24 | 23 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54
Ekman 60 Faces Test [Mean (Standard Deviation); unit: units on a scale] — The Ekman-60 Faces Test is used to assesses emotion recognition using pictures. In this study, children were presented with 60 faces across 10 actors displaying six basic emotions (i.e., happiness, sadness, disgust, fear, surprise, and anger). Facial expressions are displayed on the computer for five seconds, after which the image disappears, and participants select from a list of emotions which best described the facial expression shown. Correct responses are summed to create a total score with a possible range from 0-60, and higher scores indicate better emotion recognition.
  units on a scale | 30.84 (10.9) | 31.34 (12.94) | 31.11 (11.93)
Social Responsiveness Scale [Mean (Standard Deviation); unit: units on a scale] — The Social Responsiveness Scale identifies social impairment in children with ASD. There are five subscales, each with items scored on a scale from 1 to 4. A total score can be computed by summing scores across subscales, including, or excluding the restricted interests and repetitive behavior subscale. In this study, response options were re-coded from a scale of 1 to 4, to 0 to 3. Scores were then summed across four subscales, excluding the restrictive and repetitive behavior subscale. Possible scores ranged from 0 to 195, with higher scores meaning a better outcome.
  units on a scale | 103.28 (28.25) | 108.69 (20.92) | 106.04 (24.68)
Childhood Joint Attention Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Childhood Joint Attention Rating Scale is used to assess joint attention in children with autism spectrum disorder. In this study, we used the asocial subscale, which consists of 14 items on a scale from 0 to 4. Scores were then summed, with a possible range from 0 to 56, and higher scores mean worse joint attention.
  units on a scale | 28.09 (10.42) | 30.28 (5.93) | 29.23 (8.37)
Peabody Picture Vocabulary Test [Mean (Standard Deviation); unit: units on a scale] — The Peabody Picture Vocabulary Test assesses receptive vocabulary. The measure consists of 228 test items, each consisting of four full-color pictures as response options on a page. For each item, the examiner says a word, and the participant responds by selecting the picture that best illustrates that word's meaning. Raw scores are then summed and reported with a population mean of 100 and standard deviation of 15, with a possible range of 20 to 160. In this study, we calculated age-based standard scores, with higher scores indicating better receptive vocabulary.
  units on a scale | 87.5 (15.41) | 86.33 (19.30) | 86.88 (17.42)

OUTCOME MEASURES:

1. Primary Outcome: Ekman-60 Faces Test
Description: The Ekman-60 Faces Test is used to assesses emotion recognition using pictures. In this study, children were presented with 60 faces across 10 actors displaying six basic emotions (i.e., happiness, sadness, disgust, fear, surprise, and anger). Facial expressions are displayed on the computer for five seconds, after which the image disappears, and participants select from a list of emotions which best described the facial expression shown. Correct responses are summed to create a total score with a possible range from 0-60, and higher scores indicate better emotion recognition.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lookware TM | Lookware TM Control Module
Number analyzed (Participants) | 25 | 29
score on a scale | 38.56 (12.66) | 32.03 (13.16)

2. Primary Outcome: Social Responsiveness Scale
Description: The Social Responsiveness Scale is used to identify social impairment in children with autism spectrum disorder. The measure consists of five subscales: social motivation; social awareness; social cognition; social communication; and restricted interests and repetitive behavior, each with items scored on a scale from 1 to 4. A total score can be computed by summing scores across subscales, including, or excluding the restricted interests and repetitive behavior subscale. In this study, response options were re-coded from a scale of 1 to 4, to 0 to 3. Scores were then summed across four subscales, excluding the restrictive and repetitive behavior subscale. Possible scores ranged from 0 to 195, with higher scores meaning a better outcome.
Time Frame: 6 Weeks
Population: Missing data were not imputed for the Social Responsiveness Scale so the analysis sample for these measures differs from the other primary outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lookware TM | Lookware TM Control Module
Number analyzed (Participants) | 25 | 26
score on a scale | 90.44 (19.93) | 96.38 (20.11)

3. Secondary Outcome: Childhood Joint Attention Rating Scale
Description: The Childhood Joint Attention Rating Scale is used to assess joint attention in children with autism spectrum disorder. In this study, we used the asocial subscale, which consists of 14 items on a scale from 0 to 4. Scores were then summed, with a possible range from 0 to 56, and higher scores meant worse joint attention.
Time Frame: 6 Weeks
Population: Missing data were not imputed for the Childhood Joint Attention Rating Scale, so the analysis sample for these measures differs from the Ekman-60 Faces Test primary outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lookware TM | Lookware TM Control Module
Number analyzed (Participants) | 24 | 26
score on a scale | 27.17 (8.05) | 28.62 (7.7)

ADVERSE EVENTS:
Time Frame: Through study completion, which was approximately 6 weeks.
Arm/Group | Lookware TM | Lookware TM Control Module
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/29
Other Adverse Events (participants affected / at risk) | 0/25 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research sites that employed the PIs agreed not to disclose the trial results without the sponsor's prior written consent.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03672344/Prot_SAP_000.pdf